CLINICAL TRIAL: NCT01774331
Title: Gamma Globulin Observations and Outcomes Database for Specific Home Infusion Evidence, Patient Care And Research Data (GOOD-SHEPARD)
Acronym: GOOD-SHEPARD
Status: Terminated | Type: Observational
Why Stopped: Sponsor Decision
Sponsor: BriovaRx Infusion Services (Industry)
Responsible Party: Sponsor
Other Study IDs: AHS1-12-001
Record Dates: First submitted 2013-01-18; First posted 2013-01-24 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Intravenous Immunoglobulin (IVIg) Therapy in a Home Infusion Setting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Immunoglobulin Therapy: Immunoglobulin Therapy

SUMMARY:
Primary:

• Demonstrate the utility of a new electronic data capture (EDC) system (CareExchange™) using infusion nurse measured physical, quality of life (QOL), respiratory, and disability assessments.

Secondary:

* Change in Intravenous Immunoglobulin (IVIg) dose effects measured outcomes.
* Change in IVIg dose and timing effects measured outcomes.
* Change in patient status is reflected in measured outcomes.
* Assess the value to physicians from infusion nurse collected outcomes data.
* Identify types of patients by response to IVIg therapy (i.e. natural or poor responders).
* Change in response rate to IVIg therapy by disease state and demographics.

DETAILED DESCRIPTION:
This is a prospective, observational evaluation of immunoglobulin (Ig) therapy in consenting adult and assenting pediatric subjects who receive infusion services from BriovaRx Infusion Services, (Formerly AxelaCare Health Solutions, LLC). Subjects meeting all inclusion criteria who have provided informed consent/assent for trial participation will have validated, physician-prescribed, and standard-of-care outcome measures recorded during normal home infusion visits. Collected data will be de-identified and aggregated into cohorts of like diagnosis for trend analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age at enrollment ≥ 7
* Sign informed consent/assented to participation
* Ability to read and write English
* Understanding of study procedures and ability to comply with study procedures for the entire length of the study
* Receiving IVIg under the discretion of the patient's treating physician in accordance with standard treatment practices
* Have been on or is between doses of IVIg under the discretion of the patient's treating physician in accordance with standard treatment practices
* Being considered to be prescribed IVIg under the discretion of the patient's treating physician in accordance with standard treatment practices
* Determined to be clinically eligible for infusion services by BriovaRx Infusion Services (Formerly AxelaCare Health Solutions, LLC.) in collaboration with the patient's prescribing physician

Exclusion Criteria:

* Children (age ≤ 6 years)
* Prisoners, and other wards of the state

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient who is aged 7 years or greater at time of enrollment; who is on Ig therapy, have been on or is between doses of Ig therapy, or is being considered to be prescribed Ig therapy; provides informed consent for participation; and who has been determined to be clinically eligible for infusion services by BriovaRx Infusion Servies (Formerly AxelaCare Health Solutions, LLC), in collaboration with the patient's prescribing physician. Subjects will be recruited from the practices of participating physicians.
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2012-11; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Analysis of collected data captured in CareExchange™ will demonstrate the ability to show and track changes in outcome data. | 5 Years

SECONDARY OUTCOMES:
Physician feedback will demonstrate that having real-time access to patient data captured during a home infusion will assist in the management of the patient's disease. | 5 Years

OTHER OUTCOMES:
Demonstration of response rate for those receiving IVIg. | 5 Years
Exhibit differences in response rate of IVIg therapy across disease states and demographics. | 5 Years
Demonstration of measured variables within patients who receive IVIg. | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Allen, MD, Principal Investigator — Northwestern University and University of Minnesota
Locations (1):
- AxelaCare Health Solutions, LLC, Lenexa, Kansas, United States